CLINICAL TRIAL: NCT07261072
Title: Comparison of the Efficacy and Safety of Topical and Subcutaneous Injection of Secukinumab in HS: A Prospective Exploratory Trial
Brief Title: Comparison of the Clinical Efficacy and Safety of Topical and Subcutaneous Injection of Secukinumab in HS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Junyou ZHENG, Principal Investigator,, Peking Union Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-KY-067
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Hidradenitis Suppurativa (HS); Hidradenitis Suppurativa (Acne Inversa); Secukinumab
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical injection (Experimental)
  Interventions: Other: Topical injection of Secukinmab
- Subcutaneous injection (Active Comparator)
  Interventions: Drug: Subcutaneous injection of Secukinumab

INTERVENTIONS:
Other: Topical injection of Secukinmab — Topical injection of Secukinmab
  Arms: Topical injection
Drug: Subcutaneous injection of Secukinumab — Subcutaneous injection of Secukinumab
  Arms: Subcutaneous injection

SUMMARY:
Secukinumab is currently approved in Europe, US and China for the treatment of moderate to severe HS as a biologic agent targeting IL-17A.Two phase III clinical trials (SUNSHINE and SUNRISE) showed that 300 mg s.c. every 2 weeks resulted in 42% to 45% of patients achieving a clinical response (HiSCR) to HS, and the efficacy was sustained through 52 weeks.However, we found in clinical practice that some HS patients present with localized lesions (small areas of involvement, affecting only 1-2 anatomic areas) that are resistant to conventional therapy, and have not yet fulfilled surgical indications, and the need for systemic biologic therapy is controversial.Such patients often experience inadequate response or slow onset of action when they receive secukinumab by routine subcutaneous injection - possibly related to inadequate drug concentration in the focal lesional area and limited local anti-inflammatory effects after systemic administration.In addition, side effects of conventional subcutaneous injection system are greater, and the application is limited in some patients, so it is necessary to explore more appropriate and safer drug delivery method for localized skin lesions.Localized HS, local injection of lesions may enhance anti-inflammatory effects while reducing systemic exposure by increasing drug concentrations at the lesion site.Therefore, exploring novel modes of administration of secukinumab has practical clinical implications based on clinical practice needs and the context of the previous literature.In summary, by exploring the efficacy and safety of local skin injection of secukinumab, this study may provide a new strategy for the treatment of limited HS with sufficient scientific rationale and significant potential benefits and manageable risks.

DETAILED DESCRIPTION:
Hidradenitis suppurativa (HS) is a chronic inflammatory skin disease characterized by recurrent painful nodules, abscesses, sinus tracts, and scarring, with a global prevalence of about 1%, occurring in apocrine gland-rich areas such as the axillae and groin. Its pathogenesis is closely related to hair follicle obstruction, dysbacteriosis and immune disorders, in which IL-17A-mediated inflammatory pathways have been demonstrated to be the core driver - IL-17A levels are significantly increased in HS lesions, which can promote neutrophil infiltration and abscess formation.

Secukinumab is currently approved in Europe, US and China for the treatment of moderate to severe HS as a biologic agent targeting IL-17A.Two phase III clinical trials (SUNSHINE and SUNRISE) showed that 300 mg s.c. every 2 weeks resulted in 42% to 45% of patients achieving a clinical response (HiSCR) to HS, and the efficacy was sustained through 52 weeks.However, we found in clinical practice that some HS patients present with localized lesions (small areas of involvement, affecting only 1-2 anatomic areas) that are resistant to conventional therapy, and have not yet fulfilled surgical indications, and the need for systemic biologic therapy is controversial.Such patients often experience inadequate response or slow onset of action when they receive secukinumab by routine subcutaneous injection - possibly related to inadequate drug concentration in the focal lesional area and limited local anti-inflammatory effects after systemic administration.In addition, side effects of conventional subcutaneous injection system are greater, and the application is limited in some patients, so it is necessary to explore more appropriate and safer drug delivery method for localized skin lesions.The successful experience of topical injection of biologics in psoriasis provides an important reference for clinical practice, such as study of nail psoriasis showed that intralesional secukinumab significantly increased local drug concentrations with 73.2% improvement in nail lesions and good safety.This suggests that for localized HS, local injection of lesions may enhance anti-inflammatory effects while reducing systemic exposure by increasing drug concentrations at the lesion site.Therefore, exploring novel modes of administration of secukinumab has practical clinical implications based on clinical practice needs and the context of the previous literature.In summary, by exploring the efficacy and safety of local skin injection of secukinumab, this study may provide a new strategy for the treatment of limited HS with sufficient scientific rationale and significant potential benefits and manageable risks.

ELIGIBILITY:
Inclusion Criteria:

1. Meet international diagnostic criteria for hidradenitis suppurativa
2. Aged ≥ 18 years
3. Disease duration ≥ 6 months and resistance to conventional therapy (no significant improvement for ≥ 3 months)
4. Lesions were confined to a single anatomical area
5. Voluntarily signed the informed consent form and was able to cooperate in all visits and examinations.

Exclusion Criteria:

1. Hypersensitivity to any component of secukinumab injection
2. With severe vital organ failure
3. With active infection or malignancy (malignancy within the past 5 years, except for basal or squamous cell carcinoma of the skin and cured)
4. Treatment with biologics, immunosuppressants, or systemic corticosteroids within the last 3 months
5. Pregnant, nursing, or planning conception during the study
6. Mental disorders or cognitive impairment that precludes understanding of study procedures
7. Participating in another clinical study and are at risk of an interaction between the study drugs
8. Other conditions assessed by the investigators as inappropriate for participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in International HS Severity Score System (IHS4) | Baseline (Day 1) and Week 24
  IHS4 score is calculated by the number of nodules (multiplied by 1) plus the number of abscesses (multiplied by 2) plus the number of draining tunnels (multiplied by 4). A total score of 3 or less signifies mild disease, 4 to 10 signifies moderate disease, and 11 or higher signifies severe disease.

SECONDARY OUTCOMES:
Proportion of patients achieving Hidradenitis Suppurativa Clinical Response (HiSCR)50 | At Week4、8、12、16、20、24
  HiSCR50 is defined as at least a 50% reduction in the total abscess and inflammatory nodule count, with no increase in abscess count and no increase in draining fistula count, relative to Baseline.
Change from baseline in pain measured by Visual analog scale (VAS) | Baseline (Day 1) and week4、8、12、16、20、24
  Visual analog scale (VAS) is a simple, 1-dimensional scale that measures pain intensity, typically represented as a 10-cm horizontal line with anchors such as "no pain" and "worst possible pain."
Change from baseline in Dermatology Life Quality Index (DLQI) Total Score | Baseline (Day 1) and week4、8、12、16、20、24
  DLQI was a simple, compact, and practical questionnaire to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. The DLQI domains include symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. The participant respond on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). The DLQI total score was derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best. A lower score (that is, negative change score) indicated improvement in the Quality of Life.
Change from baseline in white blood cell count (WBC) | Baseline (Day 1) and week4、8、12、16、20、24
  A white blood cell count test measures the number of white blood cells in a sample of blood.
Change from baseline in serum level of high-density C-reactive protein (hs-CRP) | Baseline (Day 1) and week4、8、12、16、20、24
  high-density C-reactive protein (hs-CRP), which is an acute phase protein (APP), is effective for evaluating the severity and degree of inflammation in patients with HS. A normal hs-CRP level is below 3.0 mg/L. A level between 3.1-10 mg/L is considered elevated. An hs-CRP level above 10 mg/ L is very high, more likely indicating an acute inflammatory event due to infection.
Change from baseline in erythrocyte sedimentation rate (ESR) | Baseline (Day 1) and week4、8、12、16、20、24
  ESR is an indirect acute phase reactant reflecting plasma viscosity and the presence of APP, especially fibrinogen. ESR is a marker of HS disease activity. A normal range for ESR depends on your age and sex: Males younger than 50, less than 15 millimeters per hour (<15 mm/hr); males older than 50, <20mm/hr; females younger than 50, <20mm/hr; females older than 50, <30mm/hr
Change from baseline in serum level of Interleukin-6 (IL-6) | Baseline (Day 1) and week4、8、12、16、20、24
  Level of serum IL-6 is considered as an inflammatory marker. The normal range of serum IL-6 lies between 0 to 1.8 pg/mL

OTHER OUTCOMES:
Treatment-emergent adverse events (TEAEs), treatment related adverse events (TRAEs), serious adverse events (SAEs) and other safety indicators | From baseline (Day 1) to week24
  A SAE is defined as any untoward medical occurrence that, at any dose: Results in death; Is life-threatening, Requires inpatient hospitalization or prolongation of existing hospitalization; Results in persistent disability/incapacity; Is a congenital anomaly/birth defect; Important medical events. TEAEs are defined as those AEs that have a start date on or following the first dose of study treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital for Skin Diseases, Institute of Dermatology, Chinese Academy of Medical Science and Peking Union Medical College, Nanjing, Jiangsu 210042, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Griffin N, Williams AB, Anderson S, Irving PM, Sanderson J, Desai N, Goh V. Hidradenitis suppurativa: MRI features in anogenital disease. Dis Colon Rectum. 2014 Jun;57(6):762-71. doi: 10.1097/DCR.0000000000000131. PMID 24807602
- [Result] Nguyen TV, Damiani G, Orenstein LAV, Hamzavi I, Jemec GB. Hidradenitis suppurativa: an update on epidemiology, phenotypes, diagnosis, pathogenesis, comorbidities and quality of life. J Eur Acad Dermatol Venereol. 2021 Jan;35(1):50-61. doi: 10.1111/jdv.16677. Epub 2020 Jul 16. PMID 32460374
- [Result] Zouboulis CC, Desai N, Emtestam L, Hunger RE, Ioannides D, Juhasz I, Lapins J, Matusiak L, Prens EP, Revuz J, Schneider-Burrus S, Szepietowski JC, van der Zee HH, Jemec GB. European S1 guideline for the treatment of hidradenitis suppurativa/acne inversa. J Eur Acad Dermatol Venereol. 2015 Apr;29(4):619-44. doi: 10.1111/jdv.12966. Epub 2015 Jan 30. PMID 25640693
- [Result] Zouboulis CC, Bechara FG, Fritz K, Goebeler M, Hetzer FH, Just E, Kirsten N, Kokolakis G, Kurzen H, Nikolakis G, Pinter A, Podda M, Rosinski K, Schneider-Burrus S, Taube KM, Volz T, Winkler T, Kristandt A, Presser D, Zouboulis VA. S2k guideline for the treatment of hidradenitis suppurativa / acne inversa - Short version. J Dtsch Dermatol Ges. 2024 Jun;22(6):868-889. doi: 10.1111/ddg.15412. Epub 2024 May 21. PMID 38770982
- [Result] Kimball AB, Jemec GBE, Alavi A, Reguiai Z, Gottlieb AB, Bechara FG, Paul C, Giamarellos Bourboulis EJ, Villani AP, Schwinn A, Rueff F, Pillay Ramaya L, Reich A, Lobo I, Sinclair R, Passeron T, Martorell A, Mendes-Bastos P, Kokolakis G, Becherel PA, Wozniak MB, Martinez AL, Wei X, Uhlmann L, Passera A, Keefe D, Martin R, Field C, Chen L, Vandemeulebroecke M, Ravichandran S, Muscianisi E. Secukinumab in moderate-to-severe hidradenitis suppurativa (SUNSHINE and SUNRISE): week 16 and week 52 results of two identical, multicentre, randomised, placebo-controlled, double-blind phase 3 trials. Lancet. 2023 Mar 4;401(10378):747-761. doi: 10.1016/S0140-6736(23)00022-3. Epub 2023 Feb 3. PMID 36746171
- [Result] Kimball AB, Kerdel F, Adams D, Mrowietz U, Gelfand JM, Gniadecki R, Prens EP, Schlessinger J, Zouboulis CC, van der Zee HH, Rosenfeld M, Mulani P, Gu Y, Paulson S, Okun M, Jemec GB. Adalimumab for the treatment of moderate to severe Hidradenitis suppurativa: a parallel randomized trial. Ann Intern Med. 2012 Dec 18;157(12):846-55. doi: 10.7326/0003-4819-157-12-201212180-00004. PMID 23247938
- [Result] He F, Long FY, Zhang ZQ, Xia RY, Lu Y, Yin ZQ. Intramatricial injection of anti-interleukin-17A antibody for six patients with nail psoriasis. Clin Exp Dermatol. 2022 Feb;47(2):432-433. doi: 10.1111/ced.14933. Epub 2021 Oct 5. No abstract available. PMID 34510518
- [Result] Kimball AB, Okun MM, Williams DA, Gottlieb AB, Papp KA, Zouboulis CC, Armstrong AW, Kerdel F, Gold MH, Forman SB, Korman NJ, Giamarellos-Bourboulis EJ, Crowley JJ, Lynde C, Reguiai Z, Prens EP, Alwawi E, Mostafa NM, Pinsky B, Sundaram M, Gu Y, Carlson DM, Jemec GB. Two Phase 3 Trials of Adalimumab for Hidradenitis Suppurativa. N Engl J Med. 2016 Aug 4;375(5):422-34. doi: 10.1056/NEJMoa1504370. PMID 27518661
- [Result] Roccuzzo G, Repetto F, Giordano S, Sarda C, Comes A, Dapavo P, Quaglino P, Ribero S. Anti-IL17 Secukinumab in hidradenitis suppurativa: A long-term drug survival analysis. Exp Dermatol. 2024 Jul;33(7):e15140. doi: 10.1111/exd.15140. PMID 39032087
- [Result] Sabat R, Alavi A, Wolk K, Wortsman X, McGrath B, Garg A, Szepietowski JC. Hidradenitis suppurativa. Lancet. 2025 Feb 1;405(10476):420-438. doi: 10.1016/S0140-6736(24)02475-9. Epub 2025 Jan 22. PMID 39862870
- [Result] Goldburg SR, Strober BE, Payette MJ. Hidradenitis suppurativa: Epidemiology, clinical presentation, and pathogenesis. J Am Acad Dermatol. 2020 May;82(5):1045-1058. doi: 10.1016/j.jaad.2019.08.090. Epub 2019 Oct 9. PMID 31604104